CLINICAL TRIAL: NCT04471051
Title: An Observational Cohort Trial of Outcomes and Antibody Responses Following Treatment With COVID19 Convalescent Plasma in Hospitalized COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0986
Record Dates: First submitted 2020-07-13; First posted 2020-07-14 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: COVID-19; Coronavirus; SARS-CoV-2; convalescent plasma
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- COVID19 Convalescent Plasma Treatment: Hospitalized COVID19 patients who receive COVID19 Convalescent Plasma under Expanded Access protocol NCT04372368.

SUMMARY:
This is an observational study designed to learn more about how COVID19 convalescent plasma works in patients with COVID19 compared to those patients who did not receive convalescent plasma treatment. Information about patient recovery will be collected from participants' electronic medical records to evaluate safety, clinical outcomes, and SARS-CoV2 antibody responses in patients who were treated with convalescent plasma under a separate expanded access protocol, NCT04372368.

DETAILED DESCRIPTION:
This a prospective, observational cohort trial to evaluate safety, clinical outcomes, and SARS-CoV2 antibody responses in patients who were treated with anti-SARS-CoV-2 convalescent plasma under Expanded Access protocol, NCT04372368. Hospitalized patients with acute respiratory symptoms with or without confirmed interstitial COVID-19 pneumonia will be enrolled. The investigators anticipate that a minimum of 150 eligible subjects will be enrolled to receive COVID19 convalescent plasma over the 12 month period for the FDA IND expanded access protocol, NCT04372368, to provide COVID19 convalescent serum, which is a separate treatment trial. This observational protocol will co-enroll patients in parallel with the expanded access protocol and expects to enroll approximately the same number of patients but no treatment will be provided as part of this protocol. Additionally, the investigators will use Compass data with identifiers to pull information on hospitalized control COVID19+ patients from hospital admission date 4/20 to current for comparison.

This protocol is limited to data collection using the EMR to evaluate outcomes following COVID19 convalescent plasma treatment. Patient-linked specimens will not be obtained and analyzed outside of the expanded access protocol for distribution of COVID19 convalescent plasma. For this protocol, only de-identified, discarded samples may be obtained during routine patient care. Thus, consent will only be obtained from patients/subjects for participation in data abstraction/analysis from the electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Hospitalized with COVID-19 respiratory symptoms and confirmation via COVID-19 SARS-CoV-2 RT-PCR testing.
* Patient treated with COVID19 convalescent plasma.
* Patient or surrogate designated decision maker is willing and able to provide written informed consent.

Exclusion Criteria:

* Receipt of pooled immunoglobulin in past 30 days
* Contraindication to transfusion or history of prior reactions to transfusion blood products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients treated with anti-SARS-CoV-2 convalescent plasma under the Expanded Access protocol NCT04372368. Patients with acute respiratory symptoms with or without confirmed interstitial COVID-19 pneumonia will be enrolled. This observational protocol will co-enroll patients in parallel with the expanded access protocol and expects to enroll approximately the same number of patients but no treatment will be provided as part of this protocol.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Inpatient Mortality | Hospital admission up to Day 28 or discharge
  Overall Inpatient Mortality
Requirement for mechanical ventilation | Hospital admission up to Day 28 or discharge
  Number of patients requiring mechanical ventilation
Transfer to ICU | Hospital admission up to Day 28 or discharge
  Number of patients transferred to an Intensive Care Unit (ICU)
ICU Mortality | Hospital admission up to Day 28 or discharge
ICU Length of Stay (LOS) | Hospital admission up to Day 28 or discharge
  LOS, measured in days
Hospital Mortality | Hospital admission up to Day 28 or discharge
Hospital Length of Stay (LOS) | Hospital admission up to Day 28 or discharge
  LOS, measured in days

CONTACTS AND LOCATIONS:
Overall Officials: John D Beckham, MD, Principal Investigator — University of Colorado, Denver
Locations (6):
- United States (6):
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - UCHealth Memorial Hospital North, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - UCHealth Poudre Valley Hospital, Fort Collins, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado

IPD SHARING:
Plan to Share IPD: No